CLINICAL TRIAL: NCT06687109
Title: A Prospective Total Joint Surgery Registry to Monitor Short- and Long-Term Clinical Outcomes
Status: Recruiting | Type: Observational
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, MD, Spokane Joint Replacement Center
Other Study IDs: SJRC-REG
Record Dates: First submitted 2024-03-05; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Registry Knee
  Interventions: Procedure: Total Knee Arthroplasty
- Registry Hip
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total Knee Arthroplasty
  Groups: Registry Knee
Procedure: Total Hip Arthroplasty — Total Hip Arthroplasty
  Groups: Registry Hip

SUMMARY:
The investigators propose a prospective longitudinal registry study to collect and compare preoperative and postoperative information from patients who undergo total joint arthroplasty (TJA). Outcomes will be assessed with common, routinely available patient-reported outcomes measures (PROM's) such as the HOOS Jr., Oxford score, Knee Society Score, Harris Hip Score, and other patient satisfaction and function assessments in use in Orthopedics.

DETAILED DESCRIPTION:
The investigators propose a prospective longitudinal registry study to collect and compare preoperative and postoperative information from patients who undergo total joint arthroplasty (TJA). Outcomes will be assessed with common, routinely available patient-reported outcomes measures (PROM's) such as the HOOS Jr., Oxford score, Knee Society Score, Harris Hip Score, and other patient satisfaction and function assessments in use in Orthopedics. Investigators will also record both demographic and clinical data about the subject's history of joint pain, past treatment, medical co-morbidities, and surgical procedure.

Additionally, gait analysis and standardized physical capacity testing will be included as an option. All patients undergoing hip or knee replacement with the primary investigator will be included for data collection. All procedures and treatment will follow the standard of care, and all prosthetic implants with be FDA-approved. Data will be used to evaluate the effect on both short and long-term comfort and function of patients diagnosed with hip or knee pain who undergo joint replacement. The main purpose of the study is to provide quality improvement data on the patients in the Principal Investigator's (PI's) practice currently undergoing joint surgery. This project creates a data repository to store participants' data for this and possible future research.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo TJA by the Principal Investigator

Exclusion Criteria:

* Age < 18
* Unable to speak and read English
* Prisoners or any other patients who, in the opinion of the investigator, are unlikely to return for follow-ups or unreliable in completing the assessments

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For this study, we will recruit patients who are scheduled to undergo TJA by the Principal Investigator. We will include all patients aged 18 and older. The patients must be able to speak and read English. We will not enroll prisoners or any other patients who, in the opinion of the investigator, are unlikely to return for follow-ups, or would be unable to complete the PROM's. All other patients who meet eligibility criteria will be enrolled. Involvement in this study will not preclude enrollment in other studies, as the nature is non-interventional (i.e., observational).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  The Knee Society Score (KSS) provides a 0 to 100 score measuring function, pain, and range of motion in the knee before and after surgery. A score of 0 indicates the worst outcome, while a score of 100 indicates the best outcome.
Forgotten Joint Score | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  The Forgotten Joint Score assesses how aware the patient is of their joint in everyday life. A score of 0 is the worst (always aware) while a score of 100 is the best (the patient is so comfortable, they forget that the joint was replaced).
Joint Awareness Survey | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  The Joint Awareness Survey is an abbreviated version of the Forgotten Joint Score. It also has 0 as the worst outcome and 100 as the best. We are including it to determine if it can reliably be used in place of the Forgotten Joint Score, which is longer and more burdensome for patients to fill out.
Pain Satisfaction Expectations | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  This survey assesses patients' satisfaction with their joint, their pain level, their overall function, and their need for pain medication. 0 is the worst score while 100 is the best.
PROMIS Global Health | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  This survey assesses the general health and quality of life of the patient. It is also a 0-100 point scale with 100 being best, 0 being worst, and 50 being average. Every 10 points represents one standard deviation from the mean.
Koos Jr. Knee Survey | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  This survey assesses stiffness, pain, and function of the knee. 0 is the worst score and 100 is the best.
Harris Hip | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  This survey assesses pain, deformity, and range of motion of the hip. A score of 0 indicates the worst outcome and 100 indicates the best.
Hoos Jr. | Pre-op, 6 weeks, 6 months, 1 year, 2 years, and 5 years
  This survey assesses pain and function of the hip in daily life. A score of 0 indicates the worst outcome, while a score of 100 indicates the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No